CLINICAL TRIAL: NCT03356691
Title: Effects of Complementary Spirit Therapy on Servers and Patients
Brief Title: The Evaluation Complementary Spirit Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Elida Mara Carneiro da Silva, Clinic Physiotherapist, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UFTM
Record Dates: First submitted 2017-06-04; First posted 2017-11-29 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Anxiety; Depression; Pain; Well-being; Stress
Keywords: Spiritist pass; adult; laying of hands
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain | interventions — Faith Healing; Therapeutic Touch; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigators did not know which group the patients were allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control group (No Intervention): No intervention.
- Complementary Spiritist Therapy (Experimental): Prayer, Spirit education, Spiritist "passe" and magnetized water
  Interventions: Other: Complementary Spiritist Therapy
- Prayer (Other): Prayer during 1-2 minutes
  Interventions: Other: Prayer
- Spiritist "passe" (Other): Spiritist "passe" during 5-10 minutes.
  Interventions: Other: Spiritist "passe"
- Laying on of hands with intent to heal (Placebo Comparator): laying on of hands with intent to heal during 5-10 minutes.
  Interventions: Other: laying on of hands with intent to heal
- Fluid water or magnetized water (Other): Spiritist healers laying on of hands hands on the glass of water and desire health, restoration of balance and health for the patient.
  Interventions: Other: Fluid therapy.
- Non-fluidic water (Other): individuals receive water without fluidification (no laying on of hands hands on the glass of water).
  Interventions: Other: No-fluid therapy.

INTERVENTIONS:
Other: Complementary Spiritist Therapy — Complementary Spiritist Therapy:
  1. Prayer: for 1 to 2 minutes.
  2. Spiritual education: reading and commentary of the Gospel according to Spiritism, about 7 minutes.
  3. Spiritist "passe, for 2-min.
  4. Fluid therapy.
  Other Names: Integrative medicine
  Arms: Complementary Spiritist Therapy
Other: Prayer — Individuals will receive prayer during 1 to 2 minutes.
  Arms: Prayer
Other: Spiritist "passe" — Individuals will receive Spiritist "passe" during 5 to 10 minutes.
  Arms: Spiritist "passe"
Other: laying on of hands with intent to heal — Individuals will receive laying on of hands with intent to heal during 5 to 10 minutes.
  Arms: Laying on of hands with intent to heal
Other: Fluid therapy. — Individuals will receive fluid therapy.
  Arms: Fluid water or magnetized water
Other: No-fluid therapy. — Individuals will receive no-fluid therapy.
  Arms: Non-fluidic water

SUMMARY:
Background: Complementary Spiritist Therapy (ECT) based on a range of therapeutic resources including prayer, spiritist "passe", fluidotherapy (fluidic water or magnetized water), spirit education. The aim of this study was to evaluate the effects of ECT in individuals at UFTM Hospital de Clínicas.

Methods: Randomized controlled trial, patients were randomly. Patients will then be allocated into groups:

* The group submitted to ECT (prayer, spiritual education, spiritist "passe" and fluidized water or prayer or spiritist "passe" or laying on of hands with intent to heal or laying on of hands with intent to heal or fluidized water or no-fluidized water or Control group (CG) will not be submitted to any intervention.

DETAILED DESCRIPTION:
Distribution of subjects according to the group to be worked and place of data collection:

Group to be worked:

patients hospitalized in the medical and surgical clinic, orthopedics, neurology, emergency adult , gynecology and obstetrics and employees of the clinic hospital

After randomization, participants included in the study will be allocated to one of the groups:

* The group submitted to ECT:

  1. Prayer: approximation of the person to God through words including gratitude, personal petition and intercession for others, about 2 to 3 minutes;
  2. Spiritual education: reading and commentary of the Gospel according to Spiritism for about 10 minutes;
  3. Spiritist "passe": to carry out the spiritist pass, the passers-by will be asked to position themselves in front of the bed, to place their hands on the head of the person alternating with passing their hands repeatedly on or over the person, positioned lying in the dorsal position, distance about 10 to 15 cm and apply the spiritist pass for 2 to 3 minutes. Individuals will be directed to direct the thoughts in heath during the intervention;
  4. Fluid Therapy by means of magnetized or fluidized water: you will be asked to stand in front of the table containing a tray with 20 ml water cups, to place hands on the cups wishing health and healing intentions, for approximately 2 minutes .

The total time of interventions will be about 10-15 minutes.

* The control group (CG) will not be submitted to any intervention.
* The Spiritist "passe" be submitted to Spiritist "passe": To carry out the spiritist pass, the passers-by will be asked to position themselves in front of the participant, to place their hands on the head of the person alternating with passing their hands repeatedly on or over the person, distance about 10 to 15 cm and apply the spiritist pass between 5-10 minutes. Individuals will be directed the thoughts in heath during the intervention.
* The laying on of hands with intent to heal: To carry out the volunteers, the passers-by will be asked to position themselves in front of the participant, to place their hands on the head of the person alternating with passing their hands repeatedly on or over the person, distance about 10 to 15 cm and apply the spiritist pass between 5-10 minutes. Individuals will be directed the thoughts in heath during the intervention.
* The Fluid Therapy: Fluid Therapy by means of magnetized or fluidized water: you will be asked to stand in front of the table containing a tray with water cups, to place hands on the cups wishing health and healing intentions, for approximately 10 minutes.
* The No-Fluid Therapy: individuals will receive non-fluidic water.
* The Prayer group:

After intervention blood collection will be performed and the questionnaires will be applied again.

ELIGIBILITY:
Inclusion Criteria:

* The patients with the ability to understand the questionnaires.

Exclusion Criteria:

* Patients expected to be discharged in less than 4 days
* Lowering the level of consciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety sympton. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The Depression Anxiety and Stress Scale (DASS-21). This scale is a Likert 4-point scale between 0 (not applicable to me) and 3 (applies to me a lot, or most of the time). Scores for depression, anxiety and stress are determined by summing the scores of the 21 items.

SECONDARY OUTCOMES:
change in Depression. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The HAD subscale. Each of your items can be punctuated with zero to three, composing a maximum score of 21 points for each scale.
Change in Depression sympton. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The Depression Anxiety and Stress Scale (DASS-21). This scale is a Likert 4-point scale between 0 (not applicable to me) and 3 (applies to me a lot, or most of the time). Scores for depression, anxiety and stress are determined by summing the scores of the 21 items.
Change in Tension muscle. | The instrument will be applied an average on 1 day, 2 days, 3 days, 1 week, 15 days, 2 mounths.
  The visual analog scale of tension muscle. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom) orientated from the left (worst) to the right (best).
Change in wellness subjective. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The wellness subjective scale. This scale is is composed of 21 items of evaluation of positive affect, 26 items of negative affect and satisfaction with life consists of 15 items.
Change in wellness. | The instrument will be applied an average on 1 day, 2 days, 3 days, 1 week, 15 days, 2 mounths.
  The visual analog scale of wellness. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom) orientated from the left (worst) to the right (best).
Change in hematological and immunological responses. | The instrument will be applied an average on 1 day, 2 days, 3 days, 1 week, 15 days, 2 mounths.
  Hemogram, immunoglobulin A , cortisol and Cytokine Doses.
Change in pain. | The instrument will be applied an average on 1 day, 2 days, 3 days, 1 week, 15 days, 2 mounths.
  The visual analog scale of Pain. The most simple Visual Analog Pain Scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom) orientated from the left (worst) to the right (best).
Change in blood pressure | The blood pressure will be evaluated an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  Blood pressure (mmHg) is assessed by blood pressure gauge.
Change in respiratory rate | The respiratory rate will be evaluated an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  Respiratory (ipm) rate is assessed by manual count.
Change in cardiac rate | The cardiac rate will be evaluated an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  Cardiac rate (bpm) is assessed by oximeter More Fitness.
Change in oxygen saturation | The oxygen saturation will be evaluated an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  oxygen saturation (%) is assessed by oximeter More Fitness.
Change in Heart rate variability | The heart rate variability will be assessed on 1 day.
  Heart rate variability. It is measured by electrocardiogram (ECG) or frequency meter
Change in Burnout. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  Maslach Burnout Inventory. The instrument consists of 15 questions that are subdivided into three subscales: Emotional Exhaustion (EE) (5 items); Disbelief (DE) (4 items) and Professional Efficacy (EP) (6 items). All items are evaluated on a 7-point Likert scale, ranging from 0 (never) to 6 (always).
Change in Quality of life | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  Whoqol. The instrument module consists of 26 questions (being question number 1 and 2 on general quality of life), the answers follow a Likert scale (from 1 to 5, the higher the score the better the quality of life). Apart from these two questions (1 and 2), the instrument has 24 facets which comprise 4 domains that are: PHYSICAL, PSYCHOLOGICAL, SOCIAL RELATIONS and ENVIRONMENT.
Change in Stress score. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The scale of stress. This assessment is a questionnaire that evaluates stress in four levels - alert, resistance, almost exhaustion and exhaustion. The instrument assesses the presence of symptoms and how the individual has felt in the last 24 h, in the last month and in the last 3 months. For each period of time, a set of 15 physical and emotional symptoms is evaluated for the first 2 periods and 23 symptoms are evaluated for the last period.
Change in Stress. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The Depression Anxiety and Stress Scale (DASS-21). This scale is a Likert 4-point scale between 0 (not applicable to me) and 3 (applies to me a lot, or most of the time). Scores for depression, anxiety and stress are determined by summing the scores of the 21 items.
Change in perceived anxiety. | The instrument will be applied an average on 1 day, 2 days, 3 days, 1 week, 15 days, 2 mounths.
  Visual analog scale. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom) orientated from the left (worst) to the right (best).
Change in Anxiety. | The instrument will be applied an average on 1 day, 3 days, 1 week, 15 days, 2 mounths.
  The Hospital Anxiety and Depression Scale. It has 14 items, seven of which are for evaluation of anxiety (HADS-A) and seven for depression (HADS-D). Each of your items can be punctuated with zero to three, composing a maximum score of 21 points for each scale.

CONTACTS AND LOCATIONS:
Overall Officials: Élida M Carneiro, PhD, Principal Investigator — Spiritist Medical Association of Uberaba
Locations (1):
- Élida Mara Carneiro, Uberaba, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Souza Cavalcante R, Banin VB, de Moura Ribeiro Paula NA, Daher SR, Habermann MC, Habermann F, Bravin AM, da Silva CE, de Andrade LG. Effect of the Spiritist "passe" energy therapy in reducing anxiety in volunteers: A randomized controlled trial. Complement Ther Med. 2016 Aug;27:18-24. doi: 10.1016/j.ctim.2016.05.002. Epub 2016 May 6. PMID 27515871
- [Result] Carneiro EM, Moraes GV, Terra GA. Effectiveness of Spiritist Passe (Spiritual Healing) on the Psychophysiological Parameters in Hospitalized Patients. Adv Mind Body Med. 2016 Summer;30(3):4-10. PMID 27874837
- [Result] Lucchetti G, de Oliveira RF, Goncalves JP, Ueda SM, Mimica LM, Lucchetti AL. Effect of Spiritist "passe" (Spiritual healing) on growth of bacterial cultures. Complement Ther Med. 2013 Dec;21(6):627-32. doi: 10.1016/j.ctim.2013.08.012. Epub 2013 Aug 31. PMID 24280471
- [Result] Carneiro EM, Barbosa LP, Marson JM, Terra JA Junior, Martins CJ, Modesto D, Resende LA, Borges MF. Effectiveness of Spiritist "passe" (Spiritual healing) for anxiety levels, depression, pain, muscle tension, well-being, and physiological parameters in cardiovascular inpatients: A randomized controlled trial. Complement Ther Med. 2017 Feb;30:73-78. doi: 10.1016/j.ctim.2016.11.008. Epub 2016 Nov 24. PMID 28137530
- [Derived] Carneiro EM, Tosta AM, Antonelli IBS, Soares VM, Oliveira LFA, Borges RMC, da Silva AP, Borges MF. Effect of Spiritist "Passe" on Preoperative Anxiety of Surgical Patients: A Randomized Controlled Trial, Double-Blind. J Relig Health. 2020 Aug;59(4):1728-1739. doi: 10.1007/s10943-019-00841-7. PMID 31119515